CLINICAL TRIAL: NCT06371586
Title: Neo-Sequence 2：Phase 2 Study of Neoadjuvant Chemotherapy Plus Anti-angiogenesis Therapy and Immunotherapy for Locally Advanced Diffuse Gastric Cancer
Brief Title: Neo-Sequence 2：NCT Plus Anti-angiogenesis Therapy and Immunotherapy for LADGC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC4537
Record Dates: First submitted 2024-04-14; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Gastric Cancer; Diffuse Type Carcinoma
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Neoadjuvant Chemotherapy Plus Anti-angiogenesis Therapy and Immunotherapy
  Interventions: Drug: Albumin paclitaxel+SOX+BEV+ PD-1 monoclonal antibody therapy

INTERVENTIONS:
Drug: Albumin paclitaxel+SOX+BEV+ PD-1 monoclonal antibody therapy — Albumin paclitaxel+SOX+BEV bi weekly neoadjuvant therapy for 6 cycles, with PD-1 monoclonal antibody therapy interspersed for 4 cycles. Review CT and gastroscopy every 3 cycles to evaluate the therapeutic effect. Patients who have been evaluated as effective after 6 cycles of treatment may consider surgery; Or continue the two-week regimen of albumin paclitaxel+bevacizumab for 3 cycles, while PD-1 monoclonal antibody for 2 cycles. Afterwards, the therapeutic effect will be evaluated, and surgery, radiotherapy, or maintenance medication treatment will be determined based on the therapeutic effect. Surgical patients begin adjuvant treatment 1-2 months after surgery based on the curative and pathological results of the surgery. Those who fail to evaluate during neoadjuvant therapy will undergo surgery or radiation therapy, or switch to a second-line systemic treatment plan.
  Other Names: PSBP

SUMMARY:
The regimen of Albumin paclitaxel+SOX+BEV neoadjuvant therapy lasted for 6 cycles, during which PD-1 monoclonal antibody therapy was interspersed for 4 cycles for locally advanced diffuse gastric cancer.

DETAILED DESCRIPTION:
The biweekly regimen of Albumin paclitaxel+SOX+BEV neoadjuvant therapy lasted for 6 cycles, during which PD-1 monoclonal antibody therapy was interspersed for 4 cycles. Review CT and gastroscopy every 3 cycles to evaluate the therapeutic effect. Patients who have been evaluated as effective after 6 cycles of treatment may consider surgery; Or continue the dual cycle regimen ofAlbumin paclitaxel+Bevacizumab for 3 cycles, while PD-1 monoclonal antibody for 2 cycles. Afterwards, the therapeutic effect will be evaluated, and surgery, radiotherapy, or maintenance medication treatment will be determined based on the therapeutic effect. Surgical patients begin adjuvant treatment 1-2 months after surgery based on the curative and pathological results of the surgery. Those who fail to evaluate during neoadjuvant therapy will undergo surgery or radiation therapy, or switch to a second-line systemic treatment plan.

ELIGIBILITY:
Inclusion Criteria:

1. Local advanced diffuse or mixed type gastric cancer detected by pathology and endoscopy;
2. Chest, abdomen, and pelvis enhanced CT, neck and supraclavicular ultrasound, gastroscopy, and endoscopic ultrasound were used to diagnose T3-4NanyM0 gastric cancer or gastroesophageal junction cancer (refer to AJCC staging, 8th edition);
3. Has not received any anti-tumor treatment for gastric cancer yet;
4. Age range from 18 to 75 years old;
5. ECOG score 0-1 points;
6. Liver and kidney function and blood routine meet the following conditions:

   Neutrophils>1.5G/L, Hb>90g/L, PLT>100G/L; ALT and AST<2.5ULN; TBIL<1.5 ULN; Cr<1.0ULN;
7. Left ventricular ejection fraction>60%;
8. Good compliance and ability to accept long-term follow-up;
9. Sign informed consent.

Exclusion Criteria:

1. Gastrointestinal obstruction or recurrent bleeding cannot be controlled;
2. Those who cannot swallow pills;
3. Diagnose immunodeficiency or active autoimmune diseases, have received or are currently receiving immunomodulators, systemic steroid therapy, or immunosuppressive drugs within the past two years;
4. Interstitial pneumonia;
5. Moderate to severe cirrhosis caused by any reason;
6. Uncontrollable hypertension, severe kidney disease, and significant cardiovascular and cerebrovascular diseases;
7. Active infections that require systemic treatment;
8. Previously suffered from other tumors, excluding cured skin cancer and cervical cancer in situ;
9. Internal medicine diseases that do not meet the chemotherapy criteria at the same time;
10. Pregnant and lactating patients;
11. Individuals with a history of mental illness and poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Pathological response rate | 3 year
  No residual cancer cells

SECONDARY OUTCOMES:
EFS | 3 year
  event free survival
OS | 3 year
  overall survival
R0 | 3 year
  Negative margin of incision
Safety (adverse events) and surgical complications | 3 year
  Chemotherapy side effects and surgical safety

CONTACTS AND LOCATIONS:
Overall Officials: Chunxia Du, MD, Study Chair — Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Cancer hospital，Chinese acadamy of medical sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No